CLINICAL TRIAL: NCT00418366
Title: An Open- Label, 2 Part Study to Investigate the Pharmacokinetics, Safety, and Tolerability of MK0431(Sitagliptin Phosphate) in Patients With Varying Degrees of Renal Insufficiency
Brief Title: A Study on the Effect of Kidney Disease on a Diabetes Medication (0431-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-008; 2006_562
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Renal Insufficiency; Hemodialysis
Keywords: Mild, moderate, severe renal insufficiency; End stage renal disease
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular; Kidney Failure, Chronic | interventions — Sitagliptin Phosphate; Duration of Therapy

INTERVENTIONS:
Drug: MK0431, sitagliptin phosphate / Duration of Treatment : 1 Days

SUMMARY:
A study to evaluate the effect of kidney disease, from mild to severe disease, on a diabetes medication

ELIGIBILITY:
Inclusion Criteria :

* Male and non-pregnant females with a clinical diagnosis of renal insufficiency with mild, moderate, severe or end stage renal disease on hemodialysis
* A body mass index of less than 40 kg per meter squared (body weight in kg divided by height in meters squared)
* Smokes less than 10 cigarettes/day

Exclusion Criteria :

* Patients with uncontrolled diabetes or uncontrolled congestive heart failure
* Patient has abnormal prestudy laboratory measurements including serum potassium or white blood counts
* Patient has systolic blood pressure below 100 mm Hg or above 180 mm Hg
* Patient has diastolic blood pressure less than 50 mm Hg systolic or above 100 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Determination of the pharmacokinetics of MK0431 (sitagliptin phosphate) in patients with renal insufficiency compared to healthy volunteers

SECONDARY OUTCOMES:
Safety and tolerability in patients with renal insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Bergman AJ, Cote J, Yi B, Marbury T, Swan SK, Smith W, Gottesdiener K, Wagner J, Herman GA. Effect of renal insufficiency on the pharmacokinetics of sitagliptin, a dipeptidyl peptidase-4 inhibitor. Diabetes Care. 2007 Jul;30(7):1862-4. doi: 10.2337/dc06-2545. Epub 2007 Apr 27. No abstract available. PMID 17468348